CLINICAL TRIAL: NCT00268840
Title: National Trial Phase II to Study the Combination of Gemcitabine and Docetaxel in Patients With Locally Advanced or Metastatic Pancreatic or Biliary Adenocarcinoma That Cannot be Removed by Surgery
Brief Title: The Efficacy and Safety of Gemcitabine in Combination With Docetaxel to Treat Pancreatic or Biliary Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Benedicte VOTAN, ARCAGY-GINECO
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIO PANCREAS
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Pancreatic Neoplasms; Biliary Tract Neoplasms
Keywords: Pancreas or biliary cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- unique (Experimental): Taxotère - Gemzar
  Interventions: Drug: Docetaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50 mg/m2 ou 35 mg/m² (suivant le bilan hépatique) à J1 et J15 toutes les 4 semaines
  Other Names: TAXOTERE
Drug: Gemcitabine — Gemcitabine 1200 mg/m2 à J1 et J15 toutes les 4 semaines
  Other Names: GEMZAR

SUMMARY:
The purpose of this study is to assess the efficacy of combination therapy with gemcitabine and docetaxelin in patients with locally advanced or metastatic pancreatic or biliary adenocarcinoma.

DETAILED DESCRIPTION:
Try a new drug association on this advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients must sign informed consent prior to study entry
* Patients has Karnofsky performance status of more than 50%
* No prior chemotherapy
* Histologically or cytologically confirmed adenocarcinoma of the pancreas, locally advanced or metastatic disease or biliary cancer
* No previous radiotherapy for locally advanced or metastases.
* Hematopoietic: WBC > 3000/mm2, Absolute neutrophile count > 1500/mm2, Hemoglobin > 9g/dl, Platelet count > 100 000/mm2

Exclusion Criteria:

* No intracerebral or meningeal metastases
* Pregnant
* Fertile patient must use effective contraception
* No other serious medical condition or illness that would preclude study participation
* Hepatic: Bilirubin greater than upper limit of normal(ULN) SGOT and SGPT > 3.5 times upper limit of normal(ULN) alkaline phosphatase > 6 times upper limit of normal(ULN)
* More than 30 days since prior investigational therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2001-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Clinical benefit
Progression-free survival
Overall survival
To evaluate the frequency and severity of the adverse events related to the combination of gemcitabine and docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Chauvenet Laure, MD, Study Chair — ARCAGY/ GINECO GROUP
Locations (1):
- Hôpital Hôtel Dieu, Paris, France